CLINICAL TRIAL: NCT06153303
Title: A Pilot Study of Internet-based ACT for Endometriosis and Chronic Pain
Brief Title: Internet-based ACT for Endometriosis and Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Sophia Åkerblom, Associate professor, Skane University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SkaneU3
Record Dates: First submitted 2023-10-13; First posted 2023-12-01 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Endometriosis; Chronic Pain
Keywords: endometriosis; chronic pain
MeSH Terms: conditions — Endometriosis; Chronic Pain | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Acceptance and commitment therapy
  Interventions: Behavioral: Acceptance and commitment therapy

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy — The participants will go through an active internet-based ACT treatment focused on education about endometriosis and chronic pain, value-based exposure for avoided situations, and behavior change through exercises targeting the processes mindfulness, cognitive defusion and acceptance. The treatment is delivered on a safe internet platform. Participants have planned telephone contact with their assigned psychologist 2 times during the program and can also contact their psychologist via a message system in the platform and expect answer within 48 hours.

SUMMARY:
The primary aim of this study is to investigate the effect of Internet-delivered Acceptance and commitment therapy for endometriosis and chronic pain. A pilot study (no randomization; N=10) will be conducted to test the intervention and assessment procedures. The participants will go through an active internet-based ACT treatment focused on education about endometriosis and chronic pain, value-based exposure for avoided situations, and behavior change through exercises targeting the processes mindfulness, cognitive defusion and acceptance. The treatment is delivered on a safe internet platform. Participants have planned telephone contact with their assigned psychologist 2 times during the program and can also contact their psychologist via a message system in the platform and expect answer within 48 hours.

DETAILED DESCRIPTION:
Objective The primary aim of this study is to investigate the effect of Internet-delivered Acceptance and commitment therapy (iACT)for endometriosis.

Sample size 10 participants.

Trial design All participants are offered treatment. Participants are recruited from the Pain Rehabilitation Unit and the team for endometriosis at Skåne University Hospital. The unit is a government supported, regional specialist center focused on assessment and treatment of chronic pain and related disability.

Assessments Baseline and posttreatment (2 weeks after treatment) assessments will be conducted. Self-report measures will also be collected at baseline, post-treatment as well as during a 3-month follow up.

Assessment includes:Pre-and post assessment Assessors collected demographic information and self-report measures. During the pre-assessment the Mini International Neuropsychiatric Interview 5.0 (MINI) was administered to detect the presence of other comorbid disorders and assess inclusion criteria and rule out exclusion criteria.

During treatment During treatment the treatment credibility scale was administered to assess the patients' perceptions of how credible the treatment was following the introduction of the treatment rationale and the main treatment components (included in the internet program).

Safety parameters: As a mean to monitor safety and progress participants complete self-report measures (MPI, NRS, PIPS, PCS) and a question about suicidal ideation twice during the program and the therapist can follow these scores. In addition, participants can report any adverse events during treatment, at posttreatment and follow-up assessment.

Post-treatment exit interview At the post-assessment, the assigned assessor asked participants about their satisfaction with and experience of the program, what they found helpful or unhelpful and suggestions for future improvements.

Measures were taken at baseline, 2-weeks, 3 months follow-up. Self-report measures were mailed to participants

Main statistical analysis Between-group estimates on outcome will be conducted using repeated measurements. The analyses will be conducted using intention to treat principles and post hoc comparisons.

ELIGIBILITY:
Inclusion Criteria:

* verified endometriosis
* age between 18-65 years
* were fully examined medically and had received medical treatment if indicated
* were able to be an active part of the rehabilitation process, regain functioning in different life areas and participate in treatment interventions for approximately 5 hours every week
* stable dose of medication
* able to read and write in Swedish
* had access to a smart phone or computer with internet access

Exclusion Criteria:

* had acute or severe psychiatric disorders or symptoms that warranted designation as the primary disorder (ongoing substance dependence, untreated bipolar disorder, OCD, psychotic symptoms, severe depression, PTSD)
* were actively abusing analgesic medications (including narcotics), alcohol or other drugs
* had great difficulty to harbour and handle strong emotions that could lead to emotional outbursts or self-harming behavior
* had health risks due to medical reasons;
* had social or economic difficulties or lack of social support that hindered behavior change
* current severe suicidal ideation that warranted immediate intervention (indicated by the MINI and a score of 3 to item 9 of the Patient Health Questionnaire 9-item version (PHQ9))

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain interference as measured by the Multidimensional Pain Inventory (MPI) | Baseline, mid-treatment (3 weeks), mid-treatment (5 weeks), two-week-post treatment, 3 month-follow- up
  (changes between assessments) Min= 0; Max= 6. Higher scores indicate worse interference.

SECONDARY OUTCOMES:
Psychological inflexibility as measured by the Psychological Inflexibility in Pain Scale (PIPS) | Baseline, mid-treatment (3 weeks), mid-treatment (5 weeks), two-week-post treatment, 3 month-follow- up
  (changes between assessments) (changes between assessments) Min=0; Max= 52. Higher scores indicate worse inflexibility
Anxiety and depression as measured by the Hospital Anxiety and Depression Scale (HADS) | Baseline, two-week-post treatment, 3 month-follow- up
  (changes between assessments) Min= 0; Max= 21. Higher scores indicate worse depression/anxiety.
Pain intensity as measured by the Numerical Rating Scale (NRPS) | Baseline, mid-treatment (3 weeks), mid-treatment (5 weeks), two-week-post treatment, 3 month-follow- up
  (changes between assessments) Min= 0; Max= 10. Higher scores indicate worse pain intensity.
Pain catastrophizing as measured by the Pain Catastrophizing Questionnaire (PCS) | Baseline, mid-treatment (3 weeks), mid-treatment (5 weeks), two-week-post treatment, 3 month-follow- up
  (changes between assessments) Min= 0; Max= 52. Higher scores indicate worse pain catastrophizing.
Perceived health as measured by the RAND-36 Measure of Health-Related Quality of Life (RAND-36) | Baseline, two-week-post treatment, 3 month-follow- up
  (changes between assessments)Min= 0; Max= 100. Lower scores indicate worse perceived health.
Kinesiophobia as measured by the Tampa Scale of Kinesiophobia (Tampa) | Baseline, two-week-post treatment, 3 month-follow- up
  (changes between assessments) Min= 17; Max= 68. Higher scores indicate worse kinesiophobia
Health care utilization as measured by the health-care database of Region Skåne | Baseline, 3 month-follow- up
  (changes between assessments)
Health-related quality of life as measured by the Endometriosis Health Profile (EHP-30) | Baseline, two-week-post treatment, 3 month-follow- up
  (changes between assessments) Min=0; Max= 100. Lower scores indicate better health-related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne unviersity Hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No